CLINICAL TRIAL: NCT04212767
Title: The Use of Platelet-rich Fibrin in the Management of Soft Tissue Healing and Pain in Post-extraction Sockets: a Randomized Clinical Trial
Brief Title: The Use of PRF in the Management of Soft Tissue Healing
Acronym: PRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Vittorio Moraschini Filho, Principal Investigator, Universidade Federal Fluminense
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRF1
Record Dates: First submitted 2019-12-17; First posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Dental Diseases
Keywords: Tooth extraction; Platelet-rich fibrin; Soft tissue
MeSH Terms: conditions — Stomatognathic Diseases

STUDY DESIGN:
Intervention Model Description: Prospective, parallel-arm, randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Post-extraction sockets covered with Platelet-Rich Fibrin membrane (n=16)
  Interventions: Procedure: Alveolar socket preservation with Platelet-rich fibrin
- Control Goroup (No Intervention): Post-extraction sockets left to spontaneous healing/clot and primary closure (n=16).

INTERVENTIONS:
Procedure: Alveolar socket preservation with Platelet-rich fibrin — The sockets of the test group will be filled with two platelet-rich fibrin membranes followed by suture
  Other Names: Platelet-Rich Fibrin
  Arms: Test group

SUMMARY:
The present study aimed to evaluate the clinical effect of platelet-rich fibrin to improve epithelialization and decrease postoperative pain in post extraction sockets

DETAILED DESCRIPTION:
Production of PRF membranes A venipuncture was performed, prior of performing any treatment (median basilica vein, median cubital vein, median cephalic vein). Blood was drawn into four sterile, red cover tubes (IntraSpin™, Biohorizons®, Birmingham, Alabama, USA) 10-mL tubes without anticoagulant. The tubes were immediately centrifuged at 2700 rpm for 12 min (~708g) using a vertical/ fixed angle centrifuge (IntraSpin™, Biohorizons®, Birmingham, Alabama, USA). The g-force values were referenced at the bottom of the centrifugation tubes (RCF-max). After centrifugation, each L-PRF clot was removed from the tube and separated from the red element phase at the base with pliers. Four L-PRF clots were squeezed between a sterile metal plate and a metal box to obtain L-PRF membranes, similar in size and thickness.

Surgical procedures and initial clinical measurements The participants underwent periapical radiography or computed tomography (when necessary) and clinical examination to assess the absolute need for dental extraction. The participants underwent initial periodontal treatment, including supra and subgingival scaling, plaque control, and were given oral hygiene instructions.

Before tooth extraction, participants from both groups underwent local anaesthesia with mepivacaine 2% (Mepiadre, Nova DFL, Rio de Janeiro, Brazil). All teeth were extracted using a minimally traumatic procedure. No vertical releasing incisions were performed. To avoid root and bony fractures, the molar teeth were sectioned using a multilaminated drill (Zecrya, Microdont, São Paulo, Brazil). Luxation of the teeth was performed using a periotome followed by removal using forceps. After exodontia, a rigorous inspection and curettage of the socket was performed, followed by irrigation with sterile saline solution (Linhamax, Eurofarma, Rio de Janeiro, Brazil).

The sockets of the test group were filled with two PRF membranes followed by cross suture (Mononylon Ethilon, Johnson & Johnson, NJ, USA) to stabilize the membranes (Figure 1A), while the sockets of the control group received no type of biomaterial (i.e., left to spontaneous healing).

Postoperative control It was prescribed Ibuprofen (400 mg, Advil, Pfizer, São Paulo, Brazil) every 6 h was also prescribed in case of pain. Mouthwash with chlorhexidine gluconate 0.12% (Periogard, Colgate, São Paulo, Brazil) was also prescribed twice per day for 2 weeks. Sutures were removed after 10 days.

Clinical measurements One and two weeks after extraction, an assessment of soft tissue healing around the sockets was performed using the healing index system described by Landry et al (Landry, 1985). The following parameters were used to assess the level of healing: colour of tissues; epithelialisation of wound margins; presence of bleeding on palpation; granulation; and suppuration. The level of healing was scored as very poor, poor, good, very good, or excellent.

Postoperative pain and number of consumed analgesic tablets were recorded and evaluated. To assess postoperative pain, participants were instructed to complete a 10-unit visual analog scale (VAS) in combination with a graphic rating scale. The VAS ranged from 0 (no pain) to 100 (worst pain imaginable). Questionnaires were collected at the one week follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥ 18 years of age;
* Participants needing molar extraction in the mandible or maxilla region.

Exclusion Criteria:

* Smokers;
* Pregnant;
* Participants with motor difficulties that impeded or hampered hygien;
* Participants with decompensated metabolic diseases;
* Participants with periodontal disease;
* Participants with history of radiotherapy or use of bisphosphonates.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of the soft tissue epithelialization speed in post-extraction sockets | 90 days
  One and two weeks after extraction, an assessment of soft tissue healing around the sockets was performed using the healing index system described by Landry et al. The following parameters were used to assess the level of healing: colour of tissues; epithelialisation of wound margins; presence of bleeding on palpation; granulation; and suppuration. The level of healing was scored as very poor, poor, good, very good, or excellent.

SECONDARY OUTCOMES:
Postoperative pain | 90 days
  The participants were instructed to complete a 10-unit visual analog scale (VAS) in combination with a graphic rating scale. The VAS ranged from 0 (no pain) to 100 (worst pain imaginable).
Number of consumed analgesic | 90 days
  Questionnaires were collected at the one week follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Vittorio Moraschini, PhD, Principal Investigator — Fluminense Federal University
Locations (1):
- Dental Clinical Research Center of the Fluminense Federal University, Niterói, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lei L, Yu Y, Han J, Shi D, Sun W, Zhang D, Chen L. Quantification of growth factors in advanced platelet-rich fibrin and concentrated growth factors and their clinical efficacy as adjunctive to the GTR procedure in periodontal intrabony defects. J Periodontol. 2020 Apr;91(4):462-472. doi: 10.1002/JPER.19-0290. Epub 2019 Nov 17. PMID 31471902
- [Background] Castro AB, Cortellini S, Temmerman A, Li X, Pinto N, Teughels W, Quirynen M. Characterization of the Leukocyte- and Platelet-Rich Fibrin Block: Release of Growth Factors, Cellular Content, and Structure. Int J Oral Maxillofac Implants. 2019 July/August;34(4):855-864. doi: 10.11607/jomi.7275. Epub 2019 Feb 11. PMID 30742137
- [Result] Dohan DM, Choukroun J, Diss A, Dohan SL, Dohan AJ, Mouhyi J, Gogly B. Platelet-rich fibrin (PRF): a second-generation platelet concentrate. Part II: platelet-related biologic features. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Mar;101(3):e45-50. doi: 10.1016/j.tripleo.2005.07.009. Epub 2006 Jan 10. PMID 16504850